CLINICAL TRIAL: NCT07086677
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN STUDY TO DESCRIBE THE SAFETY AND TOLERABILITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE IN ADULTS
Brief Title: A Study to Learn About How a New Pneumococcal Vaccine Works in Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C4931020
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Streptococcus Pneumoniae
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (12):
- PG4 vaccine with low dose adjuvant PA-001; dose schedule 1 (Experimental)
  Interventions: Biological: PG4 vaccine in Buffer 1 with low dose PA-001
- PG4 vaccine with low dose adjuvant PA-001; dose schedule 2 (Experimental)
  Interventions: Biological: PG4 vaccine in Buffer 1 with low dose PA-001
- PG4 vaccine with low dose adjuvant PA-002; dose schedule 1 (Experimental)
  Interventions: Biological: PG4 in Buffer 1 with low dose PA-002
- PG4 vaccine with low dose adjuvant PA-002; dose schedule 2 (Experimental)
  Interventions: Biological: PG4 in Buffer 1 with low dose PA-002
- PG4 vaccine with high dose adjuvant PA-001; dose schedule 1 (Experimental)
  Interventions: Biological: PG4 in Buffer 1 with high dose PA-001
- PG4 vaccine with high dose adjuvant PA-001; dose schedule 2 (Experimental)
  Interventions: Biological: PG4 in Buffer 1 with high dose PA-001
- PG4 vaccine with high dose adjuvant PA-002; dose schedule 1 (Experimental)
  Interventions: Biological: PG4 vaccine in Buffer 1 with high dose PA-002
- PG4 vaccine with high dose adjuvant PA-002; dose schedule 2 (Experimental)
  Interventions: Biological: PG4 vaccine in Buffer 1 with high dose PA-002
- PG4 vaccine; dose schedule 1 (Active Comparator)
  Interventions: Biological: PG4 vaccine in Buffer 2; Biological: Saline injection
- PG4 vaccine; dose schedule 2 (Active Comparator)
  Interventions: Biological: PG4 vaccine in Buffer 2; Biological: Saline injection
- 20vPnC; dose schedule 1 (Active Comparator)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine; Biological: Saline injection
- 20vPnC; dose schedule 2 (Active Comparator)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine; Biological: Saline injection

INTERVENTIONS:
Biological: PG4 vaccine in Buffer 1 with low dose PA-001 — Multivalent pneumococcal conjugate vaccine
  Arms: PG4 vaccine with low dose adjuvant PA-001; dose schedule 1; PG4 vaccine with low dose adjuvant PA-001; dose schedule 2
Biological: PG4 in Buffer 1 with low dose PA-002 — Multivalent pneumococcal conjugate vaccine
  Arms: PG4 vaccine with low dose adjuvant PA-002; dose schedule 1; PG4 vaccine with low dose adjuvant PA-002; dose schedule 2
Biological: PG4 in Buffer 1 with high dose PA-001 — Multivalent pneumococcal conjugate vaccine
  Arms: PG4 vaccine with high dose adjuvant PA-001; dose schedule 1; PG4 vaccine with high dose adjuvant PA-001; dose schedule 2
Biological: PG4 vaccine in Buffer 1 with high dose PA-002 — Multivalent pneumococcal conjugate vaccine
  Arms: PG4 vaccine with high dose adjuvant PA-002; dose schedule 1; PG4 vaccine with high dose adjuvant PA-002; dose schedule 2
Biological: PG4 vaccine in Buffer 2 — Multivalent pneumococcal conjugate vaccine
  Arms: PG4 vaccine; dose schedule 1; PG4 vaccine; dose schedule 2
Biological: 20-valent pneumococcal conjugate vaccine — (20vPnC)
  Arms: 20vPnC; dose schedule 1; 20vPnC; dose schedule 2
Biological: Saline injection — Placebo
  Arms: 20vPnC; dose schedule 1; 20vPnC; dose schedule 2; PG4 vaccine; dose schedule 1; PG4 vaccine; dose schedule 2

SUMMARY:
The purpose of this study is to learn about the safety and tolerability of a pneumococcal vaccine in adults.

Participants will receive either:

* an experimental PG4 vaccine
* a PG4 vaccine comparator
* a standard 20vPnC vaccine comparator
* placebo. A placebo does not have any medicine in it but looks just like the study medicine.

Participants will take part in this study for up to 18 months depending on which group they are assigned to. During this time, the participants will receive up to two doses of study vaccine or comparator and take part in follow-up visits.

At these clinic visits, participants will be asked if any side effects were experienced. The participants will also have to give blood samples during clinic visits.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Participants either with no history of ever receiving a pneumococcal vaccine or who have received a pneumococcal vaccine more than 5 years prior to vaccination in this study

Key Exclusion Criteria:

• Participants with a history of microbiologically proven invasive disease caused by S pneumoniae.

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2027-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants reporting prespecified local reactions after each dose. | Within 7 days after each study intervention.
  Prespecified local reactions (redness, swelling, and pain at the injection site) occurring within 7 days of each dose administered in the study.
Percentage of participants reporting prespecified systemic reactions after each dose. | Within 7 days after each study intervention.
  Prespecified systemic reactions (fever, vomiting, diarrhea, headache, fatigue, muscle pain, and joint pain) occurring within 7 days of each dose administered in the study.
Percentage of participants reporting adverse events. | From signing of the ICD to 1 month after last study intervention.
  Adverse Events (AEs) occurring from Dose 1 through 1 month after the last vaccination
Percentage of participants reporting serious adverse events. | From signing of the ICD to 6 months after the last study intervention.
  Serious Adverse Events (SAEs) occurring from Dose 1 through 6 months after the last vaccination.
Percentage of participants reporting serious adverse events. | From signing of the ICD to 12 months after the last study intervention.
  Serious Adverse Events (SAEs) occurring from Dose 1 through 12 months after the last vaccination.
Percentage of participants with abnormal hematology and chemistry laboratory values. | Within 2 weeks after each study intervention.
  Any abnormal hematology or chemistry laboratory values as compared to baseline within 2 weeks after each study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Orange County Research Center, Lake Forest, California
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - CTI Clinical Research Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4931020